CLINICAL TRIAL: NCT02968095
Title: Text Message Support to Prevent Smoking Relapse in Community Treatment Settings
Brief Title: Text Message Support to Prevent Smoking Relapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miami University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23DA037320 (NIH); K23DA037320 (NIH)
Record Dates: First submitted 2016-11-15; First posted 2016-11-18 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text Message Craving Program (Experimental): Text messages designed to help smokers to modify their thinking styles to be more adaptive, delivered 2-3 times per day.
  Interventions: Behavioral: Text Message Craving Program
- Self-Help Manual Plus Control Texts (Active Comparator): A print, self-help manual plus general motivational text messages delivered 2-3 times per day.
  Interventions: Behavioral: Self-Help Manual Plus Control Texts

INTERVENTIONS:
Behavioral: Text Message Craving Program — Text messages targeting cravings delivered 2-3 times per day.
  Arms: Text Message Craving Program
Behavioral: Self-Help Manual Plus Control Texts — Self-help manual plus motivational text messages delivered 2-3 times per day.
  Arms: Self-Help Manual Plus Control Texts

SUMMARY:
The purpose of this research is to test a text message intervention for people who are beginning an attempt to quit smoking. The intervention seeks to teach people to think about their cravings to smoke in more helpful ways. The investigators expect that participants receiving the text message craving program will be less likely to begin smoking again compared to participants in a control condition.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Current daily smoking defined as smoking ≥5 cigarettes per day and having smoked for at least 3 months. During the first visit smoking status will be verified by a Carbon Monoxide level of at least 8 parts per million.
* Have a mobile phone and use text messaging at least monthly
* Be planning to quit smoking without pharmacological help.

Exclusion Criteria:

* Significant cognitive impairment
* Current therapy or pharmacological intervention for smoking or nicotine cravings
* Inability to read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
7-Day Point Prevalence Abstinence | End of Treatment (6-week) Follow-Up
  Point prevalence abstinence is defined as the prevalence of not experiencing a full relapse in the period immediately preceding measurement. A full relapse will be defined as 7 continuous days of smoking or smoking ≥ 1 day(s) per week for the two consecutive weeks preceding the time of measurement. Self-reported abstinence will be verified by a Carbon Monoxide assay of breath samples and will override self-report in the direction of smoking.

CONTACTS AND LOCATIONS:
Locations (1):
- Miami University, Oxford, Ohio, United States

IPD SHARING:
Plan to Share IPD: No